CLINICAL TRIAL: NCT06875531
Title: The Effect of Creative Drama Education on Student Nurses' Professional Nursing Value Perceptions: A Randomized Controlled Study
Brief Title: Perceptions of Student Nurses About Professional Nursing Values of Creative Drama Education
Acronym: Creative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Ebru Sevinç, Lecturer, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/25
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Creative Drama; Nurse's Role
Keywords: Creative Drama; Nursing; Perception; Education

STUDY DESIGN:
Intervention Model Description: The study will be conducted with 68 women, 34 controls and 34 interventions.
Who Masked: Participant
Masking Description: 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Content of the Training to be given Creative drama and traditional education method will consist of 5 stages. These stages are preparation, warm-up, game, improvisation, formation and evaluation stages. It is aimed to achieve the following gains by planning creative drama and traditional education in accordance with these stages for each of the concepts of human dignity, responsibility, mobilisation, safety and autonomy, which are among the professional values of the nursing profession to be addressed in the study.
  Human Dignity Outcomes Responsibility Outcomes Taking Action Outcomes Security Outcomes Autonomy Outcomes
  The experimental group will be trained with the creative drama method and the control group will be trained with the traditional teaching method in line with the learning objectives for the topics of human dignity, responsibility, mobilisation, security, autonomy.
  Interventions: Other: Creative Drama trainings
- No Intervention (No Intervention): No intervention will be made to the students in the control group after the pre-test application, and the Professional Values of Nurses Scale (HPVS) will be applied within the scope of the post-test application.
  The training given to the intervention group will be applied to the students in the control group after the post-test application.

INTERVENTIONS:
Other: Creative Drama trainings — * The experimental group will be trained with the creative drama method and the control group will be trained with the traditional teaching method in line with the learning objectives on the topics of human dignity, responsibility, taking action, safety, autonomy.
  * Creative Drama trainings will be carried out by the creative drama leader and the trainings will be continued in line with the creative drama training steps, starting with the warm-up phase, and continuing with the game, activity, improvisation and evaluation phases. Creative drama methods will be used in accordance with each topic. For each stage of the training, students will be divided into equal groups so that group members will change. Each session of creative drama training; 10 minutes for the warm-up stage, 30 minutes for the game activity stage, 30 minutes for the improvisation stage, 20 minutes for the formation and evaluation stages, and each topic will be carried out for a total of 90 minutes.
  Arms: Experimental

SUMMARY:
Objective: This study will be carried out as a pre-test-post-test randomised controlled study to examine the effect of creative drama training on the perception of professional values in nursing students.

Materials and Methods: In the study, it was planned to collect data using Personal Information Form and Professional Values of Nurses Scale (HPVS) as data collection tools. SPSS 25.0 (Statistical Package for Social Science) programme will be used for data analysis.

Design: Randomised controlled.

Study Group: The study was planned to be conducted with student nurses studying at Istanbul Arel University, Faculty of Health Sciences, Department of Nursing. The sample size of the study was calculated as a minimum of 68, 34 in the experimental group and 34 in the control group, based on Cohen's standardised effect size of 0.80 and with a power of 0.90 with the 'G. Power-3.1.9.4' programme.

DETAILED DESCRIPTION:
Professional values serve as a guide for actions accepted by professional groups and experts, providing a framework for assessing the values and beliefs that affect professional performance. For the nursing profession to achieve professional status and provide more qualified and effective care to individuals and, consequently, society, it is crucial for nurses to have a strong professional identity and professional values.

The quality of education and training plays a significant role in the development of professional professionalism. The acquisition of a professional identity begins during education and continues throughout a person's career. Therefore, creating awareness of the profession among nursing students during their student years will contribute significantly to the professionalization of the field in the future. It is essential for those who will pursue a nursing career to acquire professional values starting from their student years and to positively develop these values.

Research Question: Does the creative drama method have an effect on nursing students' perceptions of professional values (human dignity, responsibility, initiative, safety, autonomy) compared to the traditional teaching method?

ELIGIBILITY:
Inclusion Criteria:

* To have taken and successfully completed the Basic Concepts in Nursing course,
* To be registered in the Department of Nursing,
* Clinical Practice in Health Institutions,
* Volunteering to participate in the study,
* To know, understand and be able to speak Turkish

Exclusion Criteria:

-

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 5 minutes
  It consists of 8 questions including the student's age, gender, marital status, whether he/she has children, whether he/she works in another job, the number of siblings, the perception of the income status of the person, and whether there is a health worker in the family.

SECONDARY OUTCOMES:
Nurses' Professional Values Scale (HPVS) | 15 minute
  The developed scale consists of 44 items and is a five-dimensional and five-point Likert-type measurement tool. Turkish adaptation of the scale was made. The Turkish version of the scale has 36 items and the internal consistency coefficient was found to be 0.95. In this study, the total internal consistency value of the scale was found to be 0.91. The scale consists of five dimensions: human dignity, responsibility, mobilisation, security and autonomy, and the total score of the scale is calculated by averaging the scores of 36 items. The higher the mean score, the more importance nurses attach to their professional values.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Sevinç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No